CLINICAL TRIAL: NCT01540747
Title: Role of Melatonin Supplementation in Follicular Fluid of in Vitro Fertilization (IVF) Patients With Polycystic Ovarian Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Mel_FF
Record Dates: First submitted 2012-02-17; First posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2009-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: intrafollicular melatonin; PCOS; embryos quality; oocytes quality
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; Folic Acid; Melatonin

ARMS (2):
- Inofolic plus (Experimental): 178 patients
  Interventions: Dietary Supplement: Myo-inositol + folic acid + melatonin
- Inofolic (Active Comparator): 180 patients
  Interventions: Dietary Supplement: Myo-inositol + folic acid

INTERVENTIONS:
Dietary Supplement: Myo-inositol + folic acid + melatonin — Myo-inositol (2000mg)+ folic acid (200 mcg)+ melatonin(3 mg)
  Arms: Inofolic plus
Dietary Supplement: Myo-inositol + folic acid — Myo-inositol (2000mg) + folic acid (200 mcg)
  Arms: Inofolic

SUMMARY:
To evaluate the effects of melatonin supplementation on the main in vitro fertilization (IVF) outcomes during ovarian stimulation in patients with Polycystic ovarian syndrome (PCOS).

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is a common endocrine disorder that causes infertility due to anovulation in women of reproductive age. Anovulation and also decreased oocyte and embryo quality may be cause of infertility in women with PCOS. Furthermore, the reactive oxygen species (ROS) induce oxidative stress which may be responsible for poor oocyte quality. The ROS generation from mononuclear cells is elevated in women with PCOS and a significant increment of lipid peroxidation products in women with PCOS has been reported.

Melatonin is a documented powerful free radical scavenger and a broad spectrum antioxidant. It has been observed that a non-PCOS group co-treated with inositol, folic acid, and melatonin (Inofolic Plus by LO.LI.Pharma) results in a significantly greater mean number of mature oocytes, and a lower mean number of immature oocytes in patients with low oocyte quality history when compared to treatment only with inositol and folic acid (Inofolic by LO.LI.Pharma).

The aim of the study is to evaluate the possible effects of melatonin supplementation on the main IVF outcomes during ovarian stimulation of patients with PCOS.

From July 2009 to December 2011, 358 patients with PCOS (Rotterdam criteria) were enrolled in this prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PCOS
* irregular menstrual cycle (> than 28-30 days)
* normal uterine cavity
* body mass index of 20 to 26 Kg/m2
* first IVF treatment

Exclusion Criteria:

* presence of tubal, uterine, genetics and male causes of infertility
* diagnosis of cancer
* hormonal treatment in the last six months

Ages: 27 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Number of mature oocytes
embryo quality
Pregnancy rate
Implantation rate

SECONDARY OUTCOMES:
Total dose of FSH administered
Number of days of stimulation
Serum estradiol levels
Endometrial thickness
  Endometrial thickness on the day of human chorionic gonadotropin (hCG) administration
Cancellation rate
Incidence of moderate or severe ovaric hyperstimulation syndrome (OHSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Praxi Pro Vita Centro di Fertilità, Rome, Italy